CLINICAL TRIAL: NCT04453566
Title: Effect of COVID-19 Pandemic on Perceived Stress, Anxiety, Mood, and Training Quality in Elite Athletes.
Status: Completed | Type: Observational
Sponsor: Uskudar University (Other)
Collaborators: New York Medical College (Other)
Responsible Party: Principal Investigator, Ihsan Balkaya, Medical Doctor, Uskudar University
Other Study IDs: 61351342/ 2020-286
Record Dates: First submitted 2020-06-29; First posted 2020-07-01 (Actual); Last update posted 2021-04-30 (Actual); Status verified 2021-04

CONDITIONS: COVID-19; Life Satisfaction; Anxiety; Mental Health Wellness 1; Athlete; Stress
Keywords: COVID-19; Athlete; Mental Health
MeSH Terms: conditions — COVID-19; Personal Satisfaction; Anxiety Disorders; Psychological Well-Being

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Elite Athletes: Elite Athletes
  Interventions: Other: Online Survey

INTERVENTIONS:
Other: Online Survey — Online Survey

SUMMARY:
In this study, the investigator aims to measure stress, anxiety, mood, life satisfaction measures among elite athletes during COVID-19 and measure the relationship between these measures and the changes in training characteristics in elite athletes during the COVID-19 pandemic.

DETAILED DESCRIPTION:
On 11 March 2020, the World Health Organization declared the COVID-19 outbreak as a pandemic. On the same day, the first COVID-19 case reported in Turkey and nationwide quarantine regulations started after a spike in case numbers. In the world of sports, the effects of the COVID-19 pandemic started with staging games without spectators, gradually all sports events and team practices were postponed. Soon later, athletes advised to quarantine at home and continue training individually. Similar to previous study results, the COVID-19 outbreak expected to cause a profound and wide range of psychosocial impacts on people during outbreaks of infection. In fact, preliminary results from a study in China showed a moderate to severe degree psychological impact on more than half of the respondents. However, the effect of COVID-19 on mental health symptoms in elite athletes has not been investigated.

In this study, the investigator aims to investigate stress, anxiety, mood, life satisfaction measures among elite athletes during COVID-19 and explore the potential relationship between these measures and the changes in training characteristics during the COVID-19 pandemic.

ELIGIBILITY:
Inclusion Criteria:

* Elite Athletes between age of 18-35

Exclusion Criteria:

* Athletes with history of COVID-19 disease
* Athetes with first-degree family members who have/had the COVID-19 disease
* Athletes with non-covid related injuries restraining from physical activity
* History of psychiatric disease

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Elite Athletes
Sampling Method: Probability Sample
Enrollment: 208 (Actual)
Dates: Start 2020-05-27 (Actual); Primary Completion 2020-08-15 (Actual); Study Completion 2020-08-24 (Actual)

PRIMARY OUTCOMES:
Sociodemographic information and training characteristics | at inclusion
  Sociodemographic information and training characteristics Participants asked to provide sociodemographic information. Also, the difference in training frequency, duration, and quality after COVID-19 pandemic measured via 22 self-created questions.
The Beck Anxiety Inventory (BAI) | one week
  The Beck Anxiety Inventory (Beck et al., 1988) has been widely used to measure the severity of anxiety by self-report and showed to has internal consistency and high test-retest reliability. The Turkish version of the BAI proved to be a reliable and valid measure (Ulusoy et al., 1993). The participant rates how much each symptom has bothered the participant in the past week in the 21-item self-report questionnaire. The symptoms are rated on a four-point scale, ranging from ''not at all'' (0) to ''severely'' (4).
The Visual Analogue Scale (VAS) | at inclusion
  The Visual Analogue Scale (0 not stressed at all - 10 maximum amount of stress) used to measure self-reported stress and anxiety in elite athletes before and during the COVID-19 pandemic. The VAS showed to be an efficient tool for assessing self-reported stress and anxiety.
Perceived Stress Scale (PSS) | one month
  The 14-item version of PSS scale asks patients how often they had experienced thoughts and feelings such as control irritations and stress during the previous one month, with responses ranging from 0 (never) to 4 (very often). The Turkish PSS proved to be a reliable and valid tool to measure perceived stress. The final score obtained by reversing responses (e.g., 0 = 4, 1 = 3, 2 = 2, 3 = 1 & 4 = 0) to the four positively stated items (items 4, 5, 7, & 8) and then summing across all scale items. Higher scores indicating higher levels of perceived stress.
Satisfaction with Life Scale | at inclusion
  The Satisfaction with Life Scale (Diener, Emmons, Larsen, & Griffin, 1985) is a 5-item measure designed to measure global cognitive judgments of one's life satisfaction. The answers ranging from 1 (strongly disagree) to 7 (strongly agree). Items are summed to create a total score with higher scores indicating a greater degree of satisfaction with life.
Brunel mood scale (BRUMS) | at inclusion
  The BRUMs scale is based on the Profile of Mood States. The Turkish version of the BRUMS scale studied on Turkish athletes, 24-item measures and six subscales in the original version decreased to 19 items and four subscales: anger, depression, vigor, fatigue. The results of the study proved to be valid and reliable (Cakiroglu et al., 2016). Each subscale has a numerical rating scale (0 = not at all, 1 = a bit, 2 = moderate, 3 = enough; 4 = extremely) from which research participant select the one best represents at that time. The results within the subscale are summed and a score range from 0 to 16.

CONTACTS AND LOCATIONS:
Overall Officials: Mesut Karahan, PhD, Principal Investigator — Uskudar University
Locations (1):
- Uskudar University, Istanbul, Turkey (Türkiye)